CLINICAL TRIAL: NCT05749796
Title: Investigation of the Relationship Between Development, Neurological Assessment and Object Permanence in High Risk Infants.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Erkan Erol, Assistant Professor, Tokat Gaziosmanpasa University
Other Study IDs: GaziosmanpasaU_Erol_04
Record Dates: First submitted 2023-02-19; First posted 2023-03-01 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Infant Development

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study is to examine the relationship between development, neurological assessment and object permanence in risky infants aged 7-16 months. The sample of the study will consist of babies between 7-16 months at risk (preterm, low birth weight, asphyxia, hyperbillirubinemia, etc.). Inclusion criteria for the study: Between 7-16 months, having at least one risk factor. Exclusion criteria: Medical complications (eg, severe visual impairment) limiting participation in assessments; autism, down syndrome, or spinal cord injury; diagnosed uncontrolled seizure disorder; or a neurodegenerative disorder. Parents who agreed to participate in the study will be asked to fill out the demographic information questionnaire. Object permanence scale, Bayley III infant and toddler development scale and Hammersmith infant neurologic assessment will be applied to infants.

ELIGIBILITY:
Inclusion Criteria:

* Between 7-16 months, having at least one risk factor

Exclusion Criteria:

* Medical complications (eg, severe visual impairment) limiting participation in assessments; autism, down syndrome, or spinal cord injury; diagnosed uncontrolled seizure disorder; or a neurodegenerative disorder

Ages: 7 Months to 16 Months | Sex: All
Age Groups: Child
Study Population: Infants aged 7-16 months with risk factors
Sampling Method: Non-Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Object Permanence Scale | Baseline
  The minimum score of the Object Permanence Scale is 0, and the maximum score is 10. Higher scores indicate better outcome.
The Bayley Scales of Infant and Toddler Development, Third Edition (Bayley-III) motor and cognitive subscales | Baseline
  Cognitive subscale consists of 91 items and Motor subscale consists of 138 items. Items are scored as 1 (done) and 0 not able to). Higher scores indicate better outcome.
Hammersmith infant neurological assessment | Baseline
  Each item is individually scored from zero to three, and individual scores are summed to obtain a global optimality score. The overall score can range from a minimum of 0 to a maximum of 78 points.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Health Sciences, Tokat Gaziosmanpaşa University, Tokat Province, Turkey (Türkiye)